CLINICAL TRIAL: NCT00685763
Title: A Study Using Photon/Proton Beam Radiation Therapy and Chemotherapy for Unresectable Carcinoma of the Pancreas
Brief Title: Proton Therapy for Unresectable Cancer (CA) of Pancreas
Acronym: PC01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UFPTI 0609-PC01
Record Dates: First submitted 2008-05-22; First posted 2008-05-28 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic cancer; Unresectable; Proton radiation; Chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Drug Therapy; Capecitabine; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proton radiation and chemotherapy (Experimental): Chemotherapy and Radiation Combination
  Proton radiation 59.4 cobalt gray equivalent(CGE) in 33 fx at 1.8 CGE per fx over 7 weeks.
  Capecitabine (Xeloda ®) 1,000 mg by mouth approximately every 12 hrs, 5 days/week starting the first day of radiation until the end of radiation, but on radiation days only.
  Consolidation Chemotherapy starting 4 weeks after the completion of radiation
  Gemcitabine (Gemzar ®) Suggested Regimen - 1,000mg/m2 by IV over 30 minutes once a week for 3 weeks (followed by a week of rest) for 12 total doses.
  Interventions: Radiation: Proton radiation and chemotherapy

INTERVENTIONS:
Radiation: Proton radiation and chemotherapy — Proton radiation 59.4 CGE in 33 fx at 1.8 CGE per fx over 7 weeks .
  Chemotherapy:
  Capecitabine (Xeloda ®) 1,000 mg by mouth twice a day, 5 days/week (M-F) Consolidation Chemotherapy: Suggested Regimen - Gemcitabine total of 12 doses
  Other Names: Capecitabine; Xeloda; Gemcitabine; Gemzar

SUMMARY:
The purpose of this study is to find out what effects, good and/or bad, proton radiation and chemotherapy has on you and your pancreatic cancer.

DETAILED DESCRIPTION:
Chemotherapy:Capecitabine on radiation days

Proton radiation over 7 weeks

Consolidation Chemotherapy:Gemcitabine

ELIGIBILITY:
Inclusion Criteria:

Pathologically confirmed adenocarcinoma of the pancreas.

Patients must be medically inoperable or have unresectable disease

Exclusion Criteria:

* Evidence of distant metastasis; evidence of metastatic disease in the major viscera (organs), peritoneal seeding and/or ascites.
* Previous irradiation to the abdomen that would compromise the ability to deliver the prescribed treatment.
* Prior surgical resection.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-03; Primary Completion 2013-10 (Actual); Study Completion 2017-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Charles Nichols, MD, Principal Investigator — University of Florida Proton Therapy Institute
Locations (1):
- University of Florida Proton Therapy Institute, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Saif MW. Pancreatic cancer: highlights from the 42nd annual meeting of the American Society of Clinical Oncology, 2006. JOP. 2006 Jul 10;7(4):337-48. PMID 16832131
- [Background] Seydel HG, Stablein DM, Leichman LP, Kinzie JJ, Thomas PR. Hyperfractionated radiation and chemotherapy for unresectable localized adenocarcinoma of the pancreas. The Gastrointestinal Tumor Study Group experience. Cancer. 1990 Apr 1;65(7):1478-82. doi: 10.1002/1097-0142(19900401)65:73.0.co;2-3. PMID 2138054
- [Background] Schuster-Uitterhoeve AL, Gonzalez Gonzalez D, Blank LE. Radiotherapy with multiple fractions per day in pancreatic and bile duct cancer. Radiother Oncol. 1986 Nov;7(3):205-13. doi: 10.1016/s0167-8140(86)80031-7. PMID 3809584
- [Background] Ueno H, Okusaka T, Ikeda M, Tokuuye K. Phase I study of hyperfractionated radiation therapy with protracted 5-fluorouracil infusion in patients with locally advanced pancreatic cancer. Oncology. 2004;67(3-4):215-21. doi: 10.1159/000081320. PMID 15557781
- [Background] Ben-Josef E, Shields AF, Vaishampayan U, Vaitkevicius V, El-Rayes BF, McDermott P, Burmeister J, Bossenberger T, Philip PA. Intensity-modulated radiotherapy (IMRT) and concurrent capecitabine for pancreatic cancer. Int J Radiat Oncol Biol Phys. 2004 Jun 1;59(2):454-9. doi: 10.1016/j.ijrobp.2003.11.019. PMID 15145162
- [Background] Hsiung-Stripp DC, McDonough J, Masters HM, Levin WP, Hahn SM, Jones HA, Metz JM. Comparative treatment planning between proton and X-ray therapy in pancreatic cancer. Med Dosim. 2001 Fall;26(3):255-9. doi: 10.1016/s0958-3947(01)00072-3. PMID 11704461
- [Background] Mackean M, Planting A, Twelves C, Schellens J, Allman D, Osterwalder B, Reigner B, Griffin T, Kaye S, Verweij J. Phase I and pharmacologic study of intermittent twice-daily oral therapy with capecitabine in patients with advanced and/or metastatic cancer. J Clin Oncol. 1998 Sep;16(9):2977-85. doi: 10.1200/JCO.1998.16.9.2977. PMID 9738566
- [Background] Hoff PM, Ansari R, Batist G, Cox J, Kocha W, Kuperminc M, Maroun J, Walde D, Weaver C, Harrison E, Burger HU, Osterwalder B, Wong AO, Wong R. Comparison of oral capecitabine versus intravenous fluorouracil plus leucovorin as first-line treatment in 605 patients with metastatic colorectal cancer: results of a randomized phase III study. J Clin Oncol. 2001 Apr 15;19(8):2282-92. doi: 10.1200/JCO.2001.19.8.2282. PMID 11304782
- [Background] Dunst J, Reese T, Sutter T, Zuhlke H, Hinke A, Kolling-Schlebusch K, Frings S. Phase I trial evaluating the concurrent combination of radiotherapy and capecitabine in rectal cancer. J Clin Oncol. 2002 Oct 1;20(19):3983-91. doi: 10.1200/JCO.2002.02.049. PMID 12351595
- [Background] Bussels B, Goethals L, Feron M, Bielen D, Dymarkowski S, Suetens P, Haustermans K. Respiration-induced movement of the upper abdominal organs: a pitfall for the three-dimensional conformal radiation treatment of pancreatic cancer. Radiother Oncol. 2003 Jul;68(1):69-74. doi: 10.1016/s0167-8140(03)00133-6. PMID 12885454
- [Background] Eccles C, Brock KK, Bissonnette JP, Hawkins M, Dawson LA. Reproducibility of liver position using active breathing coordinator for liver cancer radiotherapy. Int J Radiat Oncol Biol Phys. 2006 Mar 1;64(3):751-9. doi: 10.1016/j.ijrobp.2005.05.066. PMID 16458774
- [Background] Korreman SS, Pedersen AN, Nottrup TJ, Specht L, Nystrom H. Breathing adapted radiotherapy for breast cancer: comparison of free breathing gating with the breath-hold technique. Radiother Oncol. 2005 Sep;76(3):311-8. doi: 10.1016/j.radonc.2005.07.009. PMID 16153728
- [Background] Sugahara S, Tokuuye K, Okumura T, Nakahara A, Saida Y, Kagei K, Ohara K, Hata M, Igaki H, Akine Y. Clinical results of proton beam therapy for cancer of the esophagus. Int J Radiat Oncol Biol Phys. 2005 Jan 1;61(1):76-84. doi: 10.1016/j.ijrobp.2004.04.003. PMID 15629597
- [Background] Bush DA, Hillebrand DJ, Slater JM, Slater JD. High-dose proton beam radiotherapy of hepatocellular carcinoma: preliminary results of a phase II trial. Gastroenterology. 2004 Nov;127(5 Suppl 1):S189-93. doi: 10.1053/j.gastro.2004.09.033. PMID 15508084
- [Background] Gierga DP, Chen GT, Kung JH, Betke M, Lombardi J, Willett CG. Quantification of respiration-induced abdominal tumor motion and its impact on IMRT dose distributions. Int J Radiat Oncol Biol Phys. 2004 Apr 1;58(5):1584-95. doi: 10.1016/j.ijrobp.2003.09.077. PMID 15050340
- [Background] Wong JW, Sharpe MB, Jaffray DA, Kini VR, Robertson JM, Stromberg JS, Martinez AA. The use of active breathing control (ABC) to reduce margin for breathing motion. Int J Radiat Oncol Biol Phys. 1999 Jul 1;44(4):911-9. doi: 10.1016/s0360-3016(99)00056-5. PMID 10386650
- [Background] Singh AK, Tierney RM, Low DA, Parikh PJ, Myerson RJ, Deasy JO, Wu CS, Pereira GC, Wahab SH, Mutic S, Grigsby PW, Hope AJ. A prospective study of differences in duodenum compared to remaining small bowel motion between radiation treatments: implications for radiation dose escalation in carcinoma of the pancreas. Radiat Oncol. 2006 Sep 4;1:33. doi: 10.1186/1748-717X-1-33. PMID 16952315
- [Background] Blackall JM, Ahmad S, Miquel ME, McClelland JR, Landau DB, Hawkes DJ. MRI-based measurements of respiratory motion variability and assessment of imaging strategies for radiotherapy planning. Phys Med Biol. 2006 Sep 7;51(17):4147-69. doi: 10.1088/0031-9155/51/17/003. Epub 2006 Aug 8. PMID 16912374
- [Background] Fishman B, Pasternak S, Wallenstein SL, Houde RW, Holland JC, Foley KM. The Memorial Pain Assessment Card. A valid instrument for the evaluation of cancer pain. Cancer. 1987 Sep 1;60(5):1151-8. doi: 10.1002/1097-0142(19870901)60:53.0.co;2-g. PMID 3300951
- [Background] Varadhachary GR, Tamm EP, Abbruzzese JL, Xiong HQ, Crane CH, Wang H, Lee JE, Pisters PW, Evans DB, Wolff RA. Borderline resectable pancreatic cancer: definitions, management, and role of preoperative therapy. Ann Surg Oncol. 2006 Aug;13(8):1035-46. doi: 10.1245/ASO.2006.08.011. Epub 2006 Jul 24. PMID 16865597
- [Background] NCCN (National Comprehensive Cancer Network) Clinical Practice Guidelines in Oncology. V.2.2006.

RESULTS

PARTICIPANT FLOW:
Groups:
- Proton Radiation and Chemotherapy: Chemotherapy and Radiation Combination
  Proton radiation 59.4 cobalt gray equivalent(CGE) in 33 fx at 1.8 CGE per fx over 7 weeks.
  Capecitabine (Xeloda ®) 1,000 mg by mouth approximately every 12 hrs, 5 days/week starting the first day of radiation until the end of radiation, but on radiation days only.
  Consolidation Chemotherapy starting 4 weeks after the completion of radiation
  Gemcitabine (Gemzar ®) Suggested Regimen - 1,000mg/m2 by IV over 30 minutes once a week for 3 weeks (followed by a week of rest) for 12 total doses.
  Proton radiation and chemotherapy: Chemotherapy Capecitabine (Xeloda ®) 1,000 mg by mouth twice a day, 5 days/week (M-F)
  Proton radiation 59.4 CGE in 33 fx at 1.8 CGE per fx over 7 weeks .
  Consolidation Chemotherapy: Suggested Regimen - Gemcitabine total of 12 doses
Period: Overall Study
Arm/Group | Proton Radiation and Chemotherapy
Started | 13
Completed | 11
Not Completed | 2
Not completed — Intercurrent death-incomplete treatment | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: Unresectable Carcinoma of the Pancreas
Groups:
- Proton Radiation and Chemotherapy: Unresectable Carcinoma of the Pancreas
Arm/Group | Proton Radiation and Chemotherapy
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: Years] | 68 [51 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of grade3+ Bowel Perforation, Grade 3+ Bleeding (Ocurring Withing 1 Years) and grade4+ Nonhematologic Acute Adverse Events (Limited to Within 90 Days of Treatment Start)
Time Frame: 1 year following the completion of radiation therapy
Measure: Number; unit: participants
Arm/Group | Proton Radiation and Chemotherapy
Number analyzed (Participants) | 11
participants | 0

2. Secondary Outcome: Collect and Analyze Tumor Control Measures
Time Frame: 1 year following the completion of radiation therapy
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year after completion of radiation therapy
Arm/Group | Proton Radiation and Chemotherapy
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Radiation and Chemotherapy (N=11)
Fatigue (General disorders) | 1 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes